CLINICAL TRIAL: NCT07258108
Title: Lucentis in Combination With Tagolimumab for the Treatment of PD-L1-Positive, HR-Positive/HER2-Negative Advanced Breast Cancer Previously Treated With CDK4/6 Inhibitors, a Phase II Study
Brief Title: Lucentis Plus Tagolimumab in PD-L1+, HR+/HER2- Advanced Breast Cancer After CDK4/6 Inhibitors
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Xu fei, Associate Chief Physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSU-2025
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lucanisatuzumab plus Tagolimumab (Experimental): Lucanisatuzumab (5 mg/kg, Q2W) in combination with tagolimumab (900 mg, Q2W) administered intraveno
  Interventions: Drug: Lucanisatuzumab plus tagolimumab

INTERVENTIONS:
Drug: Lucanisatuzumab plus tagolimumab — Each participant receives Lucanisatuzumab plus tagolimumab intravenously.

SUMMARY:
This is a Phase II single-arm study designed to evaluate the efficacy and safety of Lucanisatuzumab + Tagolisumab in 35 patients with PD-L1+ HR+/HER2- advanced breast cancer who failed prior CDK4/6 inhibitor therapy. The primary endpoint is the 6-month PFS rate. Treatment will continue until disease progression or intolerable toxicity, with periodic imaging assessments and survival follow-up.

DETAILED DESCRIPTION:
This study is a prospective, single-arm, multicenter Phase II trial designed to evaluate the efficacy and safety of Lucanisatuzumab in combination with Tagolisumab for the treatment of PD-L1-positive, HR+/HER2- advanced breast cancer patients who have failed prior CDK4/6 inhibitor therapy.

The study plans to enroll 35 patients. The primary endpoint is the 6-month progression-free survival (PFS) rate assessed by the investigator (RECIST v1.1). Secondary endpoints include PFS, objective response rate (ORR), disease control rate (DCR), duration of response (DoR), overall survival (OS), and safety. An exploratory endpoint is to analyze the correlation between TROP2 and PD-L1 expression and efficacy.

The treatment regimen consists of intravenous administration of Lucanisatuzumab (5 mg/kg, Q2W) combined with Tagolisumab (900 mg, Q2W). Treatment will continue until disease progression or occurrence of intolerable toxicity. Tumor assessments will be conducted every 6 weeks for the first 6 months, followed by every 12 weeks thereafter. Safety follow-up will occur after treatment completion, with telephone follow-ups every 3 months to collect survival and subsequent treatment information.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old.
2. HR+/HER2- breast cancer (BC), meeting the following conditions:

   1. HR+/HER2-; HER2-(IHC 0 or 1+); IHC 2+(FISH negative); HR+ (ER and/or PR IHC showed ≥1%);
   2. Tumor stage: Locally advanced, recurrent, or metastatic HR+/HER2- breast cancer; 3) Disease progression during or within 12 months after completion of adjuvant endocrine therapy based on a CDK4/6 inhibitor, or disease progression on CDK4/6 inhibitor treatment for metastatic disease; 4) PD-L1 positive (CPS ≥ 1); 5) At least one measurable target lesion as assessed by the investigator per RECIST 1.1; subjects with bone lesions only

Exclusion Criteria:

1. Received chemotherapy during the advanced stage;
2. Received any targeted therapy against topoisomerase I during the advanced stage, including antibody-drug conjugates (ADCs) (e.g., anti-CTLA-4 antibodies), immune checkpoint agonists (e.g., ICOS, CD40, CD137, GITR, OX40 antibodies), or any immune cell therapy targeting
3. Received immune checkpoint inhibitors (e.g., anti-PD-1/L1 antibodies) in the advanced stage;
4. Recurrence or metastasis within 12 months of the last chemotherapy in the early stage;
5. Subjects with central nervous system (CNS) metastases. For subjects with brain metastases who have previously received local therapy,
6. Other malignancies within 5 years prior to dosing (excluding locally treated and cured tumors such as basal cell carcinoma, squamous cell carcinoma of the skin, or cervical carcinoma in situ);

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-11-21 (Estimated); Primary Completion 2026-12-20 (Estimated); Study Completion 2026-12-26 (Estimated)

PRIMARY OUTCOMES:
progression-free survival rate (PFS) | 6 months
  The proportion of subjects who remained free of radiographic disease progression or death within 6 months of receiving the first dose of study treatment, relative to the total number of subjects.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 1 year
  The proportion of subjects achieving complete response (CR) or partial response (PR) relative to the total number of subjects
Progression-Free Survival (PFS) | 1 year
  The time from the first administration of study treatment to the first occurrence of radiographic disease progression or death, whichever occurs first
Disease Control Rate (DCR) | 1 year
  The proportion of subjects achieving complete response (CR), partial response (PR), or stable disease (SD) relative to the total number of subjects
Duration of Response (DoR) | 1 year
  The time interval from the first documented disease response to disease progression or death (whichever occurs first)
Overall survival (OS) | 1 year
  The time from the first administration of the study treatment to the participant's death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Fei Xu, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, Chile

IPD SHARING:
Plan to Share IPD: No